CLINICAL TRIAL: NCT00692536
Title: Diet Composition - Metabolic Regulation and Long-term Compliance
Acronym: KNOTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Mats Ryberg, MD, PhD, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Um dnr 07-034M
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Obesity
Keywords: Obesity; Postmenopausal; Diet intervention
MeSH Terms: conditions — Obesity | interventions — pyrophosphomevalonate decarboxylase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): NNR
  Interventions: Behavioral: NNR (Nordic Nutrition Recommendations)
- 2 (Active Comparator): MPD
  Interventions: Behavioral: MPD (Modified paleolithic diet)

INTERVENTIONS:
Behavioral: NNR (Nordic Nutrition Recommendations) — Diet with equal amounts of fat, protein and carbohydrates
  Other Names: Nordic Nutrition recommendations
  Arms: 1
Behavioral: MPD (Modified paleolithic diet) — A diet high in protein and fat, but low in carbohydrates
  Other Names: Modified paleolithic diet
  Arms: 2

SUMMARY:
This study will compare a high-protein/low-carbohydrate diet (modified paleolithic diet, MPD) with a diet high in slow carbohydrates (Nordic Nutrition Recommendations, NNR). The diets will be compared with respect effects on weight reduction, metabolic regulation, and long-term compliance to the diet regimes. Seventy-two postmenopausal overweight healthy women have been recruited and will be followed for two years.

The following variables will be studied:

* Anthropometry
* DEXA
* OGTT
* Liver fat content measured with 1H-MRS
* Hepatic 11β-HSD1 activity, measured with cortisone/cortisol conversion test

ELIGIBILITY:
Inclusion Criteria:

* Female
* Postmenopausal
* BMI>28

Exclusion Criteria:

* Disease
* Gravidity
* Smoking
* Prescribed medication

Max Age: 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Liver fat | Sept 2008

SECONDARY OUTCOMES:
Body weight | Sept 2008
Apnea-Hypopnea Index (AHI) | Sept 2008

CONTACTS AND LOCATIONS:
Overall Officials: Mats Ryberg, PhD, MD, Principal Investigator — Umeå University, Umeå, Sweden
Locations (1):
- Umeå University, Umeå, Sweden

REFERENCES:
- [Derived] Franklin KA, Lindberg E, Svensson J, Larsson C, Lindahl B, Mellberg C, Sahlin C, Olsson T, Ryberg M. Effects of a palaeolithic diet on obstructive sleep apnoea occurring in females who are overweight after menopause-a randomised controlled trial. Int J Obes (Lond). 2022 Oct;46(10):1833-1839. doi: 10.1038/s41366-022-01182-4. Epub 2022 Jul 25. PMID 35879528
- [Derived] Hooper L, Martin N, Jimoh OF, Kirk C, Foster E, Abdelhamid AS. Reduction in saturated fat intake for cardiovascular disease. Cochrane Database Syst Rev. 2020 Aug 21;8(8):CD011737. doi: 10.1002/14651858.CD011737.pub3. PMID 32827219
- [Derived] Hooper L, Martin N, Jimoh OF, Kirk C, Foster E, Abdelhamid AS. Reduction in saturated fat intake for cardiovascular disease. Cochrane Database Syst Rev. 2020 May 19;5(5):CD011737. doi: 10.1002/14651858.CD011737.pub2. PMID 32428300
- [Derived] Manousou S, Stal M, Larsson C, Mellberg C, Lindahl B, Eggertsen R, Hulthen L, Olsson T, Ryberg M, Sandberg S, Nystrom HF. A Paleolithic-type diet results in iodine deficiency: a 2-year randomized trial in postmenopausal obese women. Eur J Clin Nutr. 2018 Jan;72(1):124-129. doi: 10.1038/ejcn.2017.134. Epub 2017 Sep 13. PMID 28901333
- [Derived] Blomquist C, Alvehus M, Buren J, Ryberg M, Larsson C, Lindahl B, Mellberg C, Soderstrom I, Chorell E, Olsson T. Attenuated Low-Grade Inflammation Following Long-Term Dietary Intervention in Postmenopausal Women with Obesity. Obesity (Silver Spring). 2017 May;25(5):892-900. doi: 10.1002/oby.21815. PMID 28440046
- [Derived] Boraxbekk CJ, Stomby A, Ryberg M, Lindahl B, Larsson C, Nyberg L, Olsson T. Diet-Induced Weight Loss Alters Functional Brain Responses during an Episodic Memory Task. Obes Facts. 2015;8(4):261-72. doi: 10.1159/000437157. Epub 2015 Jul 1. PMID 26139105
- [Derived] Hammarstrom A, Wiklund AF, Lindahl B, Larsson C, Ahlgren C. Experiences of barriers and facilitators to weight-loss in a diet intervention - a qualitative study of women in northern Sweden. BMC Womens Health. 2014 Apr 16;14:59. doi: 10.1186/1472-6874-14-59. PMID 24739099